CLINICAL TRIAL: NCT00526643
Title: Gemcitabine Versus Cisplatin and Gemcitabine in First-line Treatment of Patients With Advanced Non-small Cell Lung Cancer in Poor Physical Condition (Performance Status 2)
Brief Title: CAPPA-2: Cisplatin Added to Gemcitabine in Poor Performance Advanced NSCLC Patients
Acronym: CAPPA-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: scarce enrolment and presentation of positive results of similar study in June 2012.
Sponsor: National Cancer Institute, Naples (Other)
Collaborators: Clinical Trials Promoting Group (APRIC/CTPG) (Unknown); Gruppo Oncologico del Lazio (GOL) (Unknown); Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente (Other); Gruppo Oncologico Italiano di Ricerca Clinica(GOIRC) (Unknown); Gruppo Oncologico Italia Meridionale (Other); Northwest Oncology Cooperative Group(GONO) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPPA-2; 2005-005631-97 (EudraCT Number)
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: stage IIIB; Stage IV; chemotherapy; monotherapy; combination chemotherapy; poor performance status
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm B (Experimental): combination chemotherapy
  Interventions: Drug: gemcitabine; Drug: cisplatin
- Arm A (Active Comparator): monochemotherapy
  Interventions: Drug: gemcitabine

INTERVENTIONS:
Drug: gemcitabine — 1200 mg/m2 intravenous infusion on days 1 and 8, every 3 weeks for a maximum of 4 cycles
Drug: cisplatin — cisplatin 60 mg/m2 on day 1 for 4 cycles
  Arms: Arm B

SUMMARY:
The primary objective of this study is to evaluate the impact on overall survival (OS) of the addition of cisplatin to gemcitabine vs gemcitabine alone in patients with advanced NSCLC in poor clinical condition (PS 2), not previously treated.

DETAILED DESCRIPTION:
Performance status is one of the most important prognostic factors for patients with advanced non-small cell lung cancer (NSCLC), regardless of treatment received. Chemotherapy is recommended for advanced NSCLC patients in good clinical condition, but it is not clear how much benefit is gained from giving chemotherapy to patients in poor general condition (performance status 2). This category of patients represents about 20% of all patients at initial diagnosis of NSCLC, and remains a treatment challenge for the clinician. There have been very few studies that have evaluated the impact of chemotherapy for this group of patients, and there is no established standard therapy. Studies evaluating single agent and combination two-agent chemotherapy regimens' impact on survival and improving symptoms are needed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced non small cell lung cancer, not amenable to surgical or curative radiation therapy (stage IIIB or IV);
* No prior or concomitant chemotherapy (adjuvant/neoadjuvant chemotherapy permitted if concluded at least one year prior to enrollment);
* ECOG performance status 2;
* Age: > or = 18 and < 70 years;
* Life expectancy at least 4 weeks;
* Normal bone marrow, hepatic and renal function defined as: neutrophils > or = 2000/mm3, PLT > or = 100,000/mm3, Hb > or = 10.0 g/dl, Bilirubin > or = 1.5 times the upper normal limit (UNL), AST and ALT < or = 3 times the UNL (5 times in the presence of liver metastases), creatinine within normal limits;
* Signed informed consent.

Exclusion Criteria:

* Active systemic infections;
* Severe concomitant illness (congestive heart failure, angina pectoris, myocardial infarction within previous 6 months, cardiac arrhythmias under treatment, severe arterial hypertension, severe or uncontrolled diabetes mellitus);
* Inadequate hepatic or renal function;
* Radiation therapy ongoing or concluded within two weeks prior to enrollment;
* Symptomatic cerebral metastases;
* Previous chemotherapy for advanced disease;
* Any condition that would, in the investigator's opinion, limit the patients ability to provide informed consent or to comply with study procedures;
* Pregnant or nursing females;
* Any malignancy within the past 5 years (except for adequately treated carcinoma in situ of the cervix or non melanoma skin cancer)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
overall survival | one year

SECONDARY OUTCOMES:
change in performance status | each cycle of chemotherapy
toxicity | each cycle of chemotherapy and every 3 months thereafter
quality of life | chemotherapy cycles 1 and 2
objective response | at 6 weeks and 12 weeks
progression free survival | one year

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Gridelli, M.D., Principal Investigator — APRIC/CTPG; Luciano Frontini, M.D., Principal Investigator — Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente; Vittorio Gebbia, M.D., Principal Investigator — Gruppo Oncologico Italia Meridionale; Andrea Ardizzoni, M.D., Principal Investigator — Gruppo Oncologico Italiano di Ricerca Clinica; Filippo de Marinis, M.D., Principal Investigator — GOL; Enrico Aitini, M.D., Principal Investigator — Gruppo Oncologico del Nord-Ovest; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Ciro Gallo, M.D., Ph.D., Principal Investigator — University of Campania Luigi Vanvitelli
Locations (15):
- Italy (15):
  - Azienda Ospedaliera S. Giuseppe Moscati, U.O. di Oncologia Medica, Monteforte Irpino, AV
  - Ospedale Regionale Miulli, Divisione Medicina Interna Sezione Oncologica, Acquaviva delle Fonti, BA
  - Istituto Oncologico di Bari, U.O. di Oncologia Medica e Sperimentale, Bari, BA
  - Istituto Scientifico S. Raffaele, Milan, MI
  - Azienda Ospedaliera C. Poma, Mantova, MN
  - Istituto Oncologico Veneto, Padua, PD
  - Ospedale E. Morelli, Sondalo, SO
  - Ospedale Senatore Antonio Perrino, Brindisi
  - A.O. Ospedale Mater Domini, Oncoematologia Università Magna Grecia, Catanzaro
  - Ospedale F. Veneziale, Isernia
  - A.O. Vito Fazzi, Lecce
  - Istituto Nazionale dei Tumori , Divisione di Oncologia Medica B, Napoli
  - Ospedale Regional, Unità Operative di Oncologia, Parma
  - Ospedale San Camillo - Forlanini, Rome
  - Ospedale S. Felice a Cancello, San Felice A Cancello

REFERENCES:
- [Result] Morabito A, Gebbia V, Di Maio M, Cinieri S, Vigano MG, Bianco R, Barbera S, Cavanna L, De Marinis F, Montesarchio V, Costanzo R, Sandomenico C, Montanino A, Mancuso G, Russo P, Nacci A, Giordano P, Daniele G, Piccirillo MC, Rocco G, Gridelli C, Gallo C, Perrone F. Randomized phase III trial of gemcitabine and cisplatin vs. gemcitabine alone in patients with advanced non-small cell lung cancer and a performance status of 2: the CAPPA-2 study. Lung Cancer. 2013 Jul;81(1):77-83. doi: 10.1016/j.lungcan.2013.04.008. Epub 2013 May 1. PMID 23643177
- [Derived] Gijtenbeek RG, de Jong K, Venmans BJ, van Vollenhoven FH, Ten Brinke A, Van der Wekken AJ, van Geffen WH. Best first-line therapy for people with advanced non-small cell lung cancer, performance status 2 without a targetable mutation or with an unknown mutation status. Cochrane Database Syst Rev. 2023 Jul 7;7(7):CD013382. doi: 10.1002/14651858.CD013382.pub2. PMID 37419867